CLINICAL TRIAL: NCT01825252
Title: Prevention of HIV Infection in High-Risk Social Networks of African American MSM
Brief Title: Prevention of HIV Infection in High-Risk Social Networks of African American Men Who Have Sex With Men (MSM)
Acronym: C3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Mississippi State University (Other); AIDS Task Force of Greater Cleveland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH089128 (NIH); PRO12662 (Other: Medical College of Wisconsin)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: HIV
Keywords: HIV; sexually transmitted diseases
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Network Intervention (Experimental): Approximately 20% of people in this condition will be trained to have discussions endorsing less risky behaviors with their social network members.
  Interventions: Behavioral: Social Network Intervention
- Counsel, Test, and Treat (Active Comparator): People in this arm will only receive standard-of-care counseling, testing, and treatment for HIV and STDs.
  Interventions: Behavioral: Counsel, Test, and Treat

INTERVENTIONS:
Behavioral: Social Network Intervention — Approximately 20% of people are trained to have discussions endorsing less risky behaviors with members of their social network.
  Arms: Social Network Intervention
Behavioral: Counsel, Test, and Treat — People receive standard-of-care HIV/STD counseling, testing, and treatment
  Arms: Counsel, Test, and Treat

SUMMARY:
During the formative research phase, investigators will undertake formative studies to locate, understand, and characterize high-risk social networks of African American MSM in the community; gain community participation, involvement, and input; and undertake interviews with key informants and community members to gain information needed to pilot test study recruitment procedures, measures, and intervention content.

During a 4-year main outcome trial phase, the investigators will enroll 24 separate sociocentric ("bounded") social networks composed predominantly of Black MSM. Each sociocentric network will consist of the ring of friends surrounding an initial high-risk index as well as all friends surrounding persons in this second ring and then friends surrounding a successive third snowball ring of enrollees. Each 3-ring sociocentric network is expected to consist of approximately 40 unique members (n=24 networks, each with 40 members = approximately 960 individual participants).

All participants will be assessed at baseline to measure sexual practices, substance use, and other risk characteristics over the past 3 months; asked to provide biological specimens to be tested for HIV and other sexually transmitted diseases (STDs); and counseled in HIV/STD risk reduction. STDs will be treated and those with HIV will be referred for treatment.

The investigators will identify the individuals in intervention condition networks with the greatest number of reciprocal interconnections and the most favorable sociometric standing in the network. These individuals--expected to constitute approximately 20% of the sociocentric network and designated as network leaders--will be recruited to attend a 9-session program that provides training and guidance in how to deliver on-going, theoretically-based, and culturally tailored risk reduction advice and counseling to other members within the same network.

Six and 18 months following the intervention, all participants will be reassessed on risk behavior and STD/HIV laboratory measures as well as measures of intervention exposure, with positive STD and HIV cases respectively treated or referred to care at each assessment point. Outcome analyses will test whether there is greater reduction in high-risk sexual practices, substance use associated with risky sex, and HIV/STD incidence within social networks in the intervention condition. The primary trial endpoints are reductions in prevalence and frequency of unprotected anal intercourse with nonexclusive partners, increased condom use, and lower incidence on a composite biological measure of new HIV/STD disease during the followup period.

ELIGIBILITY:
Inclusion Criteria:

* are age 18 or older;
* except for the initial index, were named as part of a friendship circle of an already-enrolled participant;
* provide written informed consent and do not exhibit intoxication, drug use,or psychiatric impairment that leads the research staff member to question capacity to provide informed consent;
* can complete study measures and participate in study activities in English;
* reside in or near the study city and do not have definite plans to leave the area in the next 12 months.

Exclusion Criteria:

* are age 17 or younger;
* exhibit intoxication, drug use, or psychiatric impairment such that they are unable to provide written informed consent;
* cannot complete study measures or adequately comprehend study activities conducted in English; or
* live in a location distant from the study city.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Actual)
Dates: Start 2011-08; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Reduction of unprotected anal intercourse with nonexclusive partners | 24 months
  We will compare the prevalence and frequency of unprotected anal intercourse with nonexclusive partners pre- and post-intervention.
Condom use | 24 months
  We will measure rates of condom pre- and post-intervention
HIV/STD incidence rates | 24 months
  We will compare HIV/STD incidence rates pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - AIDS TaskForce of Greater Cleveland, Cleveland, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Dickson-Gomez J, Owczarzak J, St Lawrence J, Sitzler C, Quinn K, Pearson B, Kelly JA, Amirkhanian YA. Beyond the ball: implications for HIV risk and prevention among the constructed families of African American men who have sex with men. AIDS Behav. 2014 Nov;18(11):2156-68. doi: 10.1007/s10461-014-0836-6. PMID 24980248
- [Background] St Lawrence JS, Kelly JA, Dickson-Gomez J, Owczarzak J, Amirkhanian YA, Sitzler C. Attitudes Toward HIV Voluntary Counseling and Testing (VCT) Among African American Men Who Have Sex With Men: Concerns Underlying Reluctance to Test. AIDS Educ Prev. 2015 Jun;27(3):195-211. doi: 10.1521/aeap.2015.27.3.195. PMID 26010312
- [Background] Quinn K, Dickson-Gomez J, DiFranceisco W, Kelly JA, St Lawrence JS, Amirkhanian YA, Broaddus M. Correlates of internalized homonegativity among black men who have sex with men. AIDS Educ Prev. 2015 Jun;27(3):212-26. doi: 10.1521/aeap.2015.27.3.212. PMID 26010313
- [Background] Broaddus MR, DiFranceisco WJ, Kelly JA, St Lawrence JS, Amirkhanian YA, Dickson-Gomez JD. Social Media Use and High-Risk Sexual Behavior Among Black Men Who Have Sex with Men: A Three-City Study. AIDS Behav. 2015 Jun;19 Suppl 2(0 2):90-7. doi: 10.1007/s10461-014-0980-z. PMID 25566762
- [Background] Kelly JA, Amirkhanian YA, Seal DW, Galletly CM, Difranceisco W, Glasman LR, Stevenson LY, Rosado N. Levels and Predictors of Sexual HIV Risk in Social Networks of Men who Have Sex with Men in the Midwest. AIDS Educ Prev. 2010 Dec;22(6):483-95. doi: 10.1521/aeap.2010.22.6.483. PMID 21204625
- [Result] Kelly JA, St Lawrence JS, Tarima SS, DiFranceisco WJ, Amirkhanian YA. Correlates of Sexual HIV Risk Among African American Men Who Have Sex With Men. Am J Public Health. 2016 Jan;106(1):96-102. doi: 10.2105/AJPH.2015.302945. Epub 2015 Nov 12. PMID 26562130
- [Result] Kelly JA, St Lawrence JS, Amirkhanian YA, DiFranceisco WJ, Anderson-Lamb M, Garcia LI, Nguyen MT. Levels and predictors of HIV risk behavior among Black men who have sex with men. AIDS Educ Prev. 2013 Feb;25(1):49-61. doi: 10.1521/aeap.2013.25.1.49. PMID 23387951
- [Result] Kelly JA, DiFranceisco WJ, St Lawrence JS, Amirkhanian YA, Anderson-Lamb M. Situational, partner, and contextual factors associated with level of risk at most recent intercourse among Black men who have sex with men. AIDS Behav. 2014 Jan;18(1):26-35. doi: 10.1007/s10461-013-0532-y. PMID 23868691